CLINICAL TRIAL: NCT00939029
Title: Highdose Nicotine Patch Therapy for Smokeless Tobacco Use
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jon Ebbert, Priniciple Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-002581; CA140125; 09-001763
Record Dates: First submitted 2009-07-10; First posted 2009-07-14 (Estimated); Results first posted 2014-04-25 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Smokeless Tobacco Use
Keywords: tobacco use; smokeless tobacco; chewing tobacco; snuff; nicotine replacement; tobacco dependence; tobacco cessation; tobacco abstinence
MeSH Terms: conditions — Tobacco Use; Tobacco Use Disorder; Tobacco Use Cessation | interventions — Nicotine Replacement Therapy; Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Active Comparator): 2 nicotine patches each at 21 mg/day for a total of 42 mg/day for 8 weeks
  Interventions: Drug: nicotine replacement therapy (nicotine patches)
- placebo (Placebo Comparator): 2 patches (containing non active ingredients) per day for 8 weeks
  Interventions: Drug: placebo NRT

INTERVENTIONS:
Drug: nicotine replacement therapy (nicotine patches) — 2- 21 mg patches per day for 8 weeks
  Arms: Active
Drug: placebo NRT — 2 placebo patches (containing no active ingredient)per day for 8 weeks
  Arms: placebo

SUMMARY:
Smokeless tobacco use ("chewing") is associated with negative health effects. To date, no medications have been shown to help chewers quit long-term. High dose nicotine patch therapy may improve the chances that chewers can quit for good. If found to be effective, chewers may use this treatment to help them quit and reduce their risk for negative health effects.

DETAILED DESCRIPTION:
Approximately 8.2 million (3.3%) of Americans ≥ 12 years of age are current smokeless tobacco (ST) users, and the prevalence of ST use has increased over the past three years. ST is increasingly being promoted as a harm reduction strategy for cigarette smoking, and two of the world's largest cigarette manufacturers have entered the ST market. ST use is estimated to be the greatest exogenous source of human exposure to cancer-causing nitrosamines. ST has been associated with oral and extra-oral cancer as well as cardiovascular and cerebrovascular mortality.

A need for efficacious interventions exists as 64% of ST users report the desire to quit. However, no pharmacotherapy has proven efficacy for increasing long-term (> 6 months) tobacco abstinence rates among ST users compared to placebo. New pharmacotherapies, drug combinations, and improved dosing of existing pharmacotherapies are needed. Previous research with nicotine patches for ST users using standard doses (up to 21 mg/day) have not increased long-term abstinence rates. However, studies of higher dose nicotine patch therapy (up to 63 mg/day) in ST users have demonstrated a dose-dependent reduction in tobacco withdrawal symptoms as well as preliminary evidence of increased long-term (> 6 months) abstinence rates compared to lower doses. The purpose of this study is to evaluate the efficacy of high dose nicotine patch therapy (42 mg/day) for increasing the 7-day point prevalence and prolonged all tobacco and ST abstinence rates at end-of-treatment (week 8), 12 and 24 weeks compared to placebo in ST users who use ≥ 3 cans/pouches per week when all subjects receive behavioral treatment for tobacco dependence. To accomplish our aims, we will randomize 60 ST users in a clinical pilot study. The work will be conducted at the Mayo Clinic in Rochester, MN.

ELIGIBILITY:
Inclusion Criteria:

1. are at least 18 years of age and at most 55 years of age;
2. report daily ST use for the past 12 months;
3. identify ST as their primary tobacco product;
4. use an average of ≥ 3 cans/pouches per week;
5. are in general good health (determined by medical history and screening physical examination);
6. have been provided with, understand, and have signed the informed consent.

Exclusion Criteria:

1. are currently using (past 30 days) any other behavioral or pharmacologic tobacco treatment program;
2. are currently pregnant or lactating;
3. have had unstable angina, myocardial infarction, or coronary angioplasty within the past 3 months;
4. have a history of arrhythmia or an abnormal tracing on the baseline EKG;
5. have a blood pressure of greater than 140/90 or a pulse of more than 110 beats per minute;
6. have a history of severe skin allergies or dermatoses;
7. have a history of intolerance to nicotine patches;
8. have another member of their household already participating in this study;
9. are taking a medication known to interact with nicotine (i.e., clozapine);
10. are taking any prescription medication for depression or asthma

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2010-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon O Ebbert, MD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Ebbert JO, Croghan IT, Schroeder DR, Hurt RD. A randomized phase II clinical trial of high-dose nicotine patch therapy for smokeless tobacco users. Nicotine Tob Res. 2013 Dec;15(12):2037-44. doi: 10.1093/ntr/ntt097. Epub 2013 Jul 19. PMID 23873976

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active | Placebo
Started | 25 | 27
Completed | 19 | 15
Not Completed | 6 | 12
Not completed — Withdrawal by Subject | 3 | 7
Not completed — Lost to Follow-up | 3 | 4
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intention to treat analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (9.1) | 35.3 (9.5) | 37.2 (9.4)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 27 | 52
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 25 | 27 | 52
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian, non-Hispanic | 23 | 26 | 49
  Caucasian, Hispanic | 2 | 1 | 3
Smokeless tobacco use [Mean (Standard Deviation); unit: cans or pouches per week] — Average cans/pouches of smokeless tobacco used per week over the last month prior to the baseline visit
  cans or pouches per week | 4.6 (1.8) | 4.0 (1.3) | 4.3 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: End of Treatment (Week 8) Point Prevalence Abstinence
Description: 7 day point prevalence abstinence at the end of treatment, biochemically confirmed by urinary anabasine < 2 ng per ml
Time Frame: weeks 8
Population: intention to treat
Measure: Number; unit: participants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 25 | 27
participants | 11 | 6
Statistical Analysis 1: Comparison: Active vs Placebo; Test type: Superiority or Other; p = 0.05, Regression, Logistic — 1 tailed p-value; Odds Ratio (OR) = 2.7, 90% CI 2-sided [1.0 to 7.5]

2. Secondary Outcome: Point-prevalence Abstinence at 3 Months
Description: 7 day point prevalence abstinence from tobacco at 3 months, biochemically confirmed using urinary anabasine < 2 ng per ml
Time Frame: week 12
Population: intention to treat
Measure: Number; unit: participants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 25 | 27
participants | 12 | 5
Statistical Analysis 1: Comparison: Active vs Placebo; Test type: Superiority or Other; p = 0.014, Regression, Logistic — 1 tailed; Odds Ratio (OR) = 4.1, 90% CI 2-sided [1.4 to 11.6]

3. Secondary Outcome: Point-prevalence Abstinence at 6 Months
Description: 7 day point prevalence abstinence from all tobacco at 6 months, biochemically confirmed using urinary anabasine < 2 ng per ml.
Time Frame: week 24
Population: intention to treat
Measure: Number; unit: participants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 25 | 27
participants | 11 | 7
Statistical Analysis 1: Comparison: Active vs Placebo; Test type: Superiority or Other; p = 0.087, Regression, Logistic — 1 tailed; Odds Ratio (OR) = 2.2, 90% CI 2-sided [0.8 to 6.0]

ADVERSE EVENTS:
Arm/Group | Active | Placebo
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/27
Other Adverse Events (participants affected / at risk) | 7/25 | 4/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=25) | Placebo (N=27)
Infection (Infections and infestations) | 1 (1) | 0 (0) — Infection was post band saw injury trauma. This occurred 4 months after subject had discontinued the patches and is not considered to be related to study drug (nicotine patches)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=25) | Placebo (N=27)
patch site reaction (Skin and subcutaneous tissue disorders) | 2 | 2
nausea (Gastrointestinal disorders) | 2 | 0
anxiety (General disorders) | 1 | 0
diarrhea (Gastrointestinal disorders) | 0 | 1
dizziness (General disorders) | 1 | 0
irritability (General disorders) | 0 | 1
itching (General disorders) | 1 | 0
sleep disturbance (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes